CLINICAL TRIAL: NCT02207972
Title: Does Ultrasound-guided CSE Technique Improve Midline Placement of Epidural Needle With Positive CSF Flow, Thereby Facilitating Correct Placement of the Catheter Compared to Catheter Placement Using Palpation of Anatomical Landmarks?
Brief Title: Does Ultrasound Help With Placement of Labor Analgesia in Pregnant Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #12-172
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy
Keywords: Pregnant; labor; Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of Ultrasound (Active Comparator): Woman requests epidural for pain relief Ultrasound guided CSE placed Continuous epidural infusion started Infusion 12 ml/hr of 0.0625% Bupivacaine and Fentanyl 2mcg/ml
  Interventions: Device: Use of Ultrasound
- No ultrasound used (Active Comparator): Palpation of anatomical landmarks Woman requests epidural for pain relief CSE placed using palpation of anatomical landmarks Continuous epidural infusion started Infusion 12 ml/hr of 0.0625% Bupivacaine and Fentanyl 2mcg/ml
  Interventions: Procedure: No ultrasound used

INTERVENTIONS:
Device: Use of Ultrasound — The ultrasound imaging of the lumbar spine in different scanning planes facilitates the identification of the landmarks necessary for appropriate epidural space location in pregnant patients. There are two acoustic windows that are effective for lumbar spine sonographic assessment: one seen on the transverse approach, and the other seen on the longitudinal paramedian approach. The ultrasound single-screen method using the transverse approach of the lumbar spine provides reliable information regarding the landmarks required for labor epidurals. The correct interspace and midline position are identified for correct placement of the CSE analgesia.
  Arms: Use of Ultrasound
Procedure: No ultrasound used — Palpation of anatomical landmarks is used for placement of labor analgesia
  Arms: No ultrasound used

SUMMARY:
The investigators believe that ultrasound guided CSE technique will accurately place the epidural needle in the midline position compared to epidural needle placement via palpation of anatomical landmarks. This will result in positive CSF in the spinal needle, correct placement of the catheter, and adequate symmetrical labor analgesia/anesthesia.

DETAILED DESCRIPTION:
Epidurals provide superior labor analgesia and anesthesia. Unfortunately, failure of epidural anesthesia and analgesia is a frequent clinical problem. In a heterogeneous cohort of 2,140 surgical patients, a failure rate of 27% for lumbar epidural was described. However, the definition of a failed epidural is broad. Different definitions include insufficient analgesia to catheter dislodgement to conversion to general anesthesia. Epidural analgesia failures may result from technical difficulties, insufficiencies or overdosing of local anesthetics, epidural septum or midline adhesions, and placement of the epidural catheter through an intervertebral foramen or into the anterior epidural space. In an imaging study of failed epidurals, incorrect catheter placement accounted for half of the failures, while the remaining patients experienced suboptimal analgesia through a correctly positioned catheter.

The incidence of overall failure was lower in patients receiving combined spinal-epidural (CSE) catheters versus epidural analgesia. In one study, the CSE technique provided decreased failure rates for labor analgesia and comparable or decreased failure rates for surgical anesthesia, when compared with reported failure rates for epidural anesthesia. It is believed that positive CSF flow in the spinal needle confirms correct epidural needle placement in the epidural space and also confirms the epidural needle to be in the midline position. Placement of the epidural needle in the midline position will minimize the incorrect placement of the catheter to one side, providing a symmetrical analgesia versus unilateral analgesia.

However, the practice of CSE and epidural catheter placement relies on the palpation of anatomical landmarks that are not always easy to feel. Therefore, the epidural needle maybe placed "off midline" despite positive loss of resistance (LOR) that causes negative CSF flow in the spinal needle and an incorrectly placed catheter. As a result, the incorrect catheter placement will result in a "failed" or suboptimal epidural analgesia.

Ultrasound has recently been utilized to facilitate lumbar epidurals and spinals. The US imaging of the lumbar spine in different scanning planes facilitates the identification of the landmarks necessary for appropriate epidural space location in pregnant patients. There are two acoustic windows that are effective for lumbar spine sonographic assessment: one seen on the transverse approach, and the other seen on the longitudinal paramedian approach. The ultrasound single-screen method using the transverse approach of the lumbar spine provides reliable information regarding the landmarks required for labor epidurals. The correct interspace and midline position are identified for correct placement of the CSE analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparious
* Term (>37 weeks gestation)
* Vertex presentation
* Singleton gestation
* Ability to provide informed consent
* Request for analgesia for labor pain
* Maternal age 18 years or greater

Exclusion Criteria:

* Multiparous
* Preterm (< 37 weeks gestation)
* Presentation other than vertex (breech, transverse)
* Active drug/alcohol dependence
* Previous spinal surgeries
* Known spinal deformities

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Migdalia Saloum, MD, Principal Investigator — Mount Sinai Roosevelt Hospital
Locations (1):
- Mount-Sinai Roosevelt hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in labor requesting epidural will be offered to participate in the study for their neuraxial placement
Pre-assignment Details: Once the patient agrees to be in the study, they will be randomized into one of the 2 arms (with or without ultrasound) for their neuraxial placement.
Period: Overall Study
Arm/Group | Use of Ultrasound | No Ultrasound Used
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Use of Ultrasound | No Ultrasound Used | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Full Range); unit: years] | 31.83 [19 to 39] | 31.85 [19 to 39] | 31.84 [19 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate Epidural Placement
Description: Number of ultrasound guided CSE technique accurately placed epidural needle in the midline position
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Groups:
- Use of Ultrasound: Woman requests epidural for pain relief Ultrasound guided CSE placed
  Continuous epidural infusion started Infusion 12 ml/hr of 0.0625% Bupivacaine and Fentanyl 2mcg/ml
  Use of Ultrasound: The ultrasound imaging of the lumbar spine in different scanning planes
Arm/Group | Use of Ultrasound | No Ultrasound Used
Number analyzed (Participants) | 22 | 24
Participants | 21 | 23

2. Secondary Outcome: Number of Participants With Successful First Attempt
Description: The number of participants who had first attempt success to locate the epidural space and midline position
Time Frame: Immediate
Population: Pregnant patients in labor requesting neuraxial analgesia
Measure: Count of Participants; unit: Participants
Arm/Group | Use of Ultrasound | No Ultrasound Used
Number analyzed (Participants) | 22 | 24
Participants | 19 | 21

3. Secondary Outcome: Number of Participants Without Angle Adjustments in Space Success
Description: the number of participants with successes without any readjustment of the angle in the space
Time Frame: immediate
Measure: Count of Participants; unit: Participants
Arm/Group | Use of Ultrasound | No Ultrasound Used
Number analyzed (Participants) | 22 | 24
Participants | 16 | 12

ADVERSE EVENTS:
Groups:
- No Ultrasound Used: Palpation of anatomical landmarks Woman requests epidural for pain relief CSE placed using palpation of anatomical landmarks
  Continuous epidural infusion started Infusion 12 ml/hr of 0.0625% Bupivacaine and Fentanyl 2mcg/ml
  No ultrasound used: Palpation of anatomical landmarks is used for placement of labor analgesia
Arm/Group | Use of Ultrasound | No Ultrasound Used
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No